CLINICAL TRIAL: NCT02111720
Title: Maybe, Maybe Not: Deciding to Disclose HIV Status to Family
Brief Title: Disclosure to Family
Acronym: D2F
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of South Florida (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MH097486; R01MH097486 (NIH)
Record Dates: First submitted 2014-03-28; First posted 2014-04-11 (Estimated); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: HIV Risk Reduction; Attention Control Case Management
Keywords: HIV; Disclosure; Family; Intervention
MeSH Terms: interventions — Calcibiotic Root Canal Sealer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Maybe, Maybe Not (Experimental): The intervention is an individual-level 4-session + 3 month booster series designed to assist persons with HIV in making decisions regarding the disclosure of their HIV serostatus to family members.
  Interventions: Behavioral: Maybe, Maybe Not
- Comprehensive Risk Counseling and Services (Active Comparator): Comprehensive Risk Counseling and Services (CRCS) will be used to provide the attention-placebo control (CDC, 2006). CRCS combines traditional case management and HIV risk-reduction in an individualized, client-centered program which focuses on the reduction of risk behavior and addresses a client's psychosocial and medical needs.
  Interventions: Behavioral: Comprehensive Risk Counseling and Services

INTERVENTIONS:
Behavioral: Maybe, Maybe Not — The goals of session one are to introduce participants to the intervention, to assess current decision context, to assist in the clarification of participant values, and to encourage the participant to set specific goals for disclosure decision-making. The goals for session two are to explore the participants' motivations to disclose or not to disclose and the potential costs and rewards of both disclosing and not disclosing. The goals for session three are to guide participants through disclosure decision making, and to support comfort/acceptance with decisions made. The goal of session four is to support the decision-making process. The booster session is used to reinforce the effects of the intervention through continued discussion of disclosure decisions in the preceding months, strategies used in disclosing, and rewards and costs of decision-making.
  Arms: Maybe, Maybe Not
Behavioral: Comprehensive Risk Counseling and Services — CRCS combines traditional case management and HIV risk-reduction in an individualized, client-centered program which focuses on the reduction of risk behavior and addresses a client's psychosocial and medical needs.CRCS focuses on seven core elements: recruitment and engagement; screening, enrolling, and assessing; prevention planning; risk reduction counseling; referrals and service coordination; monitoring; and discharge and maintenance. These core elements represent the framework of the intervention, and provide enough flexibility to allow implementation that most appropriately serves the needs of clients.
  Other Names: CRCS
  Arms: Comprehensive Risk Counseling and Services

SUMMARY:
The decision to disclose one's serostatus to family members creates considerable emotional strain for people living with HIV (PLWH), regardless of gender and sexual orientation. While disclosure to family members has been linked to positive outcomes including increased social support, improved health outcomes (i.e., sexual, physical, mental), reduced loneliness and stress, and improved HIV disease management, the decision not to disclose can also lead to positive outcomes. To date, most research about serostatus disclosure has focused on the act of disclosing - the who, what, where, and when of disclosing - rather than the decision process involved. The investigator's long-range goal is to further refine and evaluate an intervention designed to enhance HIV disclosure decision-making among PLWH. To reach this goal, the investigators are proposing a course of study with the following specific aims: Specific Aim 1. Assess the effectiveness of the intervention relative to an attention-control condition on a variety of primary outcomes related to disclosure and health. Specific Aim 2: Examine the effects of the intervention over time. Specific Aim 3: Explore the potential mediating effects of disclosure decision making on the primary outcomes. Specific Aim 4: Explore potential moderating effects of participant demographics (e.g., gender, age), relationship characteristics (i.e., relationship satisfaction, proximity, importance of disclosure), and contextual variables related to family (e.g., adaptability, problem-solving) on intervention effectiveness. Specific Aim 5: Evaluate the effects of treatment engagement, retention and expectations on outcomes.

DETAILED DESCRIPTION:
A two-armed, randomized, parallel group, attention-placebo control design is proposed to assess the relative efficacy of the intervention. Participants who meet the enrollment criteria will complete baseline assessments prior to being randomized into one of two intervention groups: the experimental group or the ACCM. The ACCM will function as a concurrent control group. All participants will receive four individualized sessions of interventional procedures, regardless of assignment. The first 3 sessions will take place at weekly intervals, with a 4-week wait period between sessions 3 and 4. The wait period permits those in the experimental arm to consider disclosure decisions, and to make disclosures if they so choose. Participants in both groups will return for assessment and a booster session at 3-months post-baseline. Participants in both groups will also return at 6- and 12-months post-baseline for follow-up assessments.

Experimental Condition is: Maybe or Maybe Not. The intervention is an individual-level 4-session + 3 month booster series designed to assist persons with HIV in making decisions regarding the disclosure of their HIV serostatus to family members. The CTD asserts that HIV-positive persons weigh the rewards and costs of disclosing their status to family. Whenever the rewards outweigh the costs, disclosure occurs. In previous work, this theory has proven to be an effective model in understanding disclosure to family and friends. The goals of session one are to introduce participants to the intervention, to assess current decision context, to assist in the clarification of participant values, and to encourage the participant to set specific goals for disclosure decision-making. Participants will explore their current family relationships, and determine which family members they want to consider telling, and which family members they know they don't want to tell. Participants are then asked to complete the disclosure decisions assessment with the facilitator. This assessment is used to gather information about the decision context specific to each family member. Participants identify each family members' disclosure status (i.e., aware/not aware), as well as other key attributes of each relationship which inform the decision such as importance of disclosure and satisfaction with the relationship. A series of handouts designed to initiate awareness of the decision process are then provided and discussed. For example, a handout entitled, "Questions to ask yourself as you think about disclosing to family members," is used to stimulate and expand awareness of the context within which disclosure decisions will be made. The goals for session two are to explore the participants' motivations to disclose or not to disclose and the potential costs and rewards of both disclosing and not disclosing. Strategies that can be employed to minimize disclosure-related costs are also reviewed. The goals for session three are to guide participants through disclosure decision making, and to support comfort/acceptance with decisions made. Only when a decision to disclose has been made, participants will complete a Family Disclosure Worksheet, to rehearse potential disclosure conversations, and to prepare for the potential reactions of family members. Where the decision is made not to disclose, emphasis is placed on supporting comfort/acceptance with this decision. Through discussions with their facilitator, participants are encouraged to consider the ongoing nature of the decision-making and evaluation processes. The goal of session four is to support the decision-making process. If applicable, the session begins with a review of the Family Disclosure Worksheet and all other intervention materials. The decision-making process is reviewed, and comfort and acceptance with each decision is again explored. Participants are encouraged to reflect on their readiness to make disclosure decisions with respect to specific family members. If the decision not to disclose is made, the session focus includes support of that decision, and a discussion of the cues for assessment and re-evaluation. Preliminary data from the pilot study suggest that disclosures were still occurring at 3-months post-intervention, indicating that a booster session may be helpful. In addition to initial exposure to "treatment," effective interventions generally include some follow-up or booster sessions to support durability of impact. Low frequency booster sessions following the termination of an intensive treatment have been proposed as one method that may assist in maintaining treatment gains, and have been shown to be effective for a variety of therapeutic interventions including behavioral family therapy, anger management, assertions skills training, behavioral psychotherapy, and HIV prevention. In this study a 3-month booster session will be used to reinforce the effects of the intervention through continued discussion of disclosure decisions in the preceding months, strategies used in disclosing, and rewards and costs of decision-making.

The Control condition is: Attention control case management (ACCM). The CDC's HIV Prevention case management program "Comprehensive Risk Counseling and Services" (CRCS) will be used to provide the attention-placebo control. CRCS combines traditional case management and HIV risk-reduction in an individualized, client-centered program which focuses on the reduction of risk behavior and addresses a client's psychosocial and medical needs. HIV-positive individuals often have numerous psychosocial, financial, and medical challenges, and may not immediately acknowledge the need for prevention services because their basic living needs (e.g., housing) are more salient. CRCS focuses on seven core elements: recruitment and engagement; screening, enrolling, and assessing; prevention planning; risk reduction counseling; referrals and service coordination; monitoring; and discharge and maintenance. These core elements represent the framework of the intervention, and provide enough flexibility to allow implementation that most appropriately serves the needs of clients. Trust is a key element in the ability to work with participants. In the ACCM, the facilitator will work in cooperation with the participant using a problem-solving approach geared to build trust, and will place emphasis on connecting the participant to community-based services and supports. As operationalized by the AIDS and Substance Abuse Program, the initial CRCS meeting provides an opportunity to describe the program, gather information and establish rapport. For those who present with immediate needs such as for shelter or medical care, this first meeting may provide an opportunity for linking the participant to services immediately. The initial treatment plan is developed in the second meeting. The facilitator will go through each of six general areas with the participant to gather a history and picture of the current situation: (1) substance abuse; (2) basic needs; (3) health care; (4) mental health; (5) legal issues; and (6) support systems. Once this review is complete, an initial intervention plan is developed with specific goals and objectives. Case management is a continual process of developing goals, working to meet those goals and addressing obstacles. Thus, the ACCM can mimic the experimental condition, and will be delivered on the same session schedule as the experimental condition and will include a comparable booster session at 3 months. Facilitators will be extensively trained by the PI and will be knowledgeable regarding local resources for HIV-positive persons. Facilitators will be qualified to make appropriate referrals to service providers and to local AIDS service organizations (ASOs), and will evaluate participant referral follow-through by encouraging a discussion of referral activities at each session. Resource lists provided to participants in both groups during the first session will include contact information for a 24-hour hotline in the event of emergency.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive men and women
* over the age of 18
* indicate an interest in learning more about disclosure
* have at least one family member who does not know of diagnosis
* sexually active in past 90 days
* speak and understand English
* plan on living in Tampa area for at least one year

Exclusion Criteria:

* not HIV-positive
* children under the age of 18
* not able to speak and understand English
* do not plan on living in Tampa area for the year
* not sexually active in last 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2013-07; Primary Completion 2020-08-17 (Estimated); Study Completion 2020-08-17 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to 52 weeks in HIV Transmission Risk | Baseline, Week 7, Week 12, Week 24, Week 52
  Ordinal measure of HIV transmission risk. The ordinal measure is constructed from information provided by the participant on the last five sexual encounters during the prior 30 days, with the highest risk assigned to encounters involving discordant anal/vaginal intercourse, unprotected, with a discordant partner (XEF)

SECONDARY OUTCOMES:
Change from baseline to 52 weeks in the number of family members to whom participants have disclosed their positive serostatus | Baseline, Week 7, Week 12, Week 24, Week 52
  At baseline, the ASSIS interview tool is used to identify participants' family members who do not know the participants' serostatus. During the study period, they will report any of these family members to whom they disclosure their serostatus (i.e., the status of disclosure has changed from "not disclosed to" to "disclosed to")
Change from baseline to 52 weeks in the odds of disclosure to sex partners | Baseline, Week 7, Week 12, Week 24, Week 52
  Participants will indicate, for each of their last 5 encounters, whether or not they disclosed their serostatus to sex partners (DPA)
Change from baseline to 52 weeks in the proportion of sex partners disclosed to | Baseline, Week 7, Week 12, Week 24, Week 52
  Participants will indicate the number of sex partners disclosed to during the prior 30 days (DBC)

OTHER OUTCOMES:
Change from baseline to 52 weeks in depression score (CES-D) | Baseline, Week 7, Week 12, Week 24, Week 52
  Participants provide depression scores on the 20-item Center for Epidemeologic Studies Depression Scale
Change from baseline to 52 weeks in anxiety score (CAS) | Baseline, Week 7, Week 12, Week 24, Week 52
  Anxiety assessed with the 9-item Costello-Comrey Anxiety Scale.
Change from baseline to 52 weeks in self-esteem score (SERS) | Baseline, Week 7, Week 12, Week 24, Week 52
  Self-esteem assessed with the 40-item Self-Esteem Rating Scale.
Change from baseline to 52 weeks in coping score (WCI) | Baseline, Week 7, Week 12, Week 24, Week 52
  Coping assessed with the 50-item Ways of Coping Inventory
Change from baseline to 52 weeks in HIV Stigma score (STG) | Baseline, Week 7, Week 12, Week 24, Week 52
  HIV Stigma assessed with the 40-item HIV Stigma scale
Change from baseline to 52 weeks in health (MDH) | Baseline, Week 7, Week 12, Week 24, Week 52
  General health and physical functioning assessed with the 21-item Multidimensional Health Scale
Change from baseline to 52 weeks in unprotected anal intercourse | Baseline, Week 7, Week 12, Week 24, Week 52
  Participants are asked to provide the number of sexual encounters involving unprotected anal intercourse during the prior 30 day period (XBC)

CONTACTS AND LOCATIONS:
Overall Officials: Julianne M Serovich, PhD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States